CLINICAL TRIAL: NCT04226300
Title: Laparoscopic-Assisted Versus Ultrasound-Guided Visualization of Transversus Abdominis Plane Blocks
Brief Title: Lap-assisted vs. US-Guided Visualization of TAP Blocks
Acronym: LUV-TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephanie D. Chao, Assistant Professor of Pediatric Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 44988
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative
Keywords: transversus abdominus plane; nerve block; TAP block; laparoscopic vs. ultrasound; post-op pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Laparoscopy; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive a TAP block either by the surgeon, laparoscopically, or by the anesthesia team via ultrasound guidance.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, their families, post-anesthesia care unit nurses and anesthesiologists reviewing images of the ultrasound will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic-Assisted (Experimental): Surgeons will place TAP block laparoscopically using a camera prior to beginning a surgical procedure.
  Interventions: Procedure: Laparoscopic
- Ultrasound-Guided (Active Comparator): Anesthesiologists will use ultrasound to place TAP block prior to beginning a surgical procedure.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Laparoscopic — A transversus abdominis nerve block will be placed laparoscopically.
  Arms: Laparoscopic-Assisted
Procedure: Ultrasound — A transversus abdominis nerve block will be place by ultrasound
  Arms: Ultrasound-Guided

SUMMARY:
Peripheral nerve blocks have been effective in decreasing post-operative pain as well as the use of narcotics for numerous years. Typically, these blocks are placed by anesthesiologist via ultrasound. In more recent years, surgeons have been placing nerve blocks laparoscopically. Since there are few studies that looks compare the two techniques we aim to perform a randomized control trial to demonstrate if a laparoscopic placed nerve block is as efficient and accurate as an ultrasound placed block.

DETAILED DESCRIPTION:
Ultrasound-guided peripheral nerve blocks like the transversus abdominis plane (TAP) block are useful for post-operative pain control and reducing opioid analgesics.(1-3) A recent meta-analysis of TAP blocks in adults demonstrated a reduction in post-operative opioid requirements, and improved pain scores.(2) Within the pediatric population, numerous other studies have confirmed the benefit of TAP blocks and their ability to lower pain scores, reduce opioid use and opioid-related side effects post-operatively.(4) While there have been many prospective randomized trials for ultrasound-guided TAP blocks (5-7), there has been limited evaluation of surgically-placed TAP blocks (8). There has been no published data evaluating or comparing surgically placed TAP blocks in pediatric patients undergoing laparoscopic procedures. placed TAP blocks in pediatrics have not been examined in patients undergoing laparoscopic procedures.(4) Our pilot study was designed as a proof of concept, to demonstrate that ultrasound images could be used to verify the distribution of local anesthetic after a laparoscopically-assisted TAP block. The aim of this study is to continue using ultrasound to verify the location of laparoscopic-assisted TAP blocks, and compare the post-operative outcomes (pain scores, opioid use, etc.) to those who receive ultrasound-guided TAP blocks. We plan to do this in a prospective, randomized and semi-blinded fashion.

We hypothesize that (1) we will be able to accurately describe the location of the TAP block placed by both methods in more than 90% of cases; (2) laparoscopic-assisted TAP blocks will be as effective as ultrasound-guided TAP blocks in terms of managing/reducing post-operative pain scores and reducing the amount and frequency of postoperative opioid analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 0-18 years who are undergoing laparoscopic surgery at Lucille Packard Children's Hospital
* Clinical indication for abdominal peripheral nerve block

Exclusion Criteria:

* conversion to open procedure
* allergy to local anesthetic
* multiple procedures planned with >1 surgical specialty

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Transversus abdominis plane (TAP) block location | 2 years
  Images of the TAP block will be taken and reviewed by anesthesiologists to document the location of the block
Post-operative pain | 24 hours
  The Face Pain Scale (Hicks et. al., 2001) is a self-reported scale that uses cartoon depictions of faces to quantify on a scale 0-10 scale how pain a child is experiencing at a given moment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Chao, MD, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. PMID 21154380
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Petersen PL, Mathiesen O, Torup H, Dahl JB. The transversus abdominis plane block: a valuable option for postoperative analgesia? A topical review. Acta Anaesthesiol Scand. 2010 May;54(5):529-35. doi: 10.1111/j.1399-6576.2010.02215.x. Epub 2010 Feb 17. PMID 20175754
- [Background] Mai CL, Young MJ, Quraishi SA. Clinical implications of the transversus abdominis plane block in pediatric anesthesia. Paediatr Anaesth. 2012 Sep;22(9):831-40. doi: 10.1111/j.1460-9592.2012.03916.x. PMID 22834467
- [Background] Carney J, Finnerty O, Rauf J, Curley G, McDonnell JG, Laffey JG. Ipsilateral transversus abdominis plane block provides effective analgesia after appendectomy in children: a randomized controlled trial. Anesth Analg. 2010 Oct;111(4):998-1003. doi: 10.1213/ANE.0b013e3181ee7bba. Epub 2010 Aug 27. PMID 20802056
- [Background] Sandeman DJ, Bennett M, Dilley AV, Perczuk A, Lim S, Kelly KJ. Ultrasound-guided transversus abdominis plane blocks for laparoscopic appendicectomy in children: a prospective randomized trial. Br J Anaesth. 2011 Jun;106(6):882-6. doi: 10.1093/bja/aer069. Epub 2011 Apr 18. PMID 21504934
- [Background] Fredrickson MJ, Paine C, Hamill J. Improved analgesia with the ilioinguinal block compared to the transversus abdominis plane block after pediatric inguinal surgery: a prospective randomized trial. Paediatr Anaesth. 2010 Nov;20(11):1022-7. doi: 10.1111/j.1460-9592.2010.03432.x. PMID 20964768
- [Background] Ravichandran NT, Sistla SC, Kundra P, Ali SM, Dhanapal B, Galidevara I. Laparoscopic-assisted Tranversus Abdominis Plane (TAP) Block Versus Ultrasonography-guided Transversus Abdominis Plane Block in Postlaparoscopic Cholecystectomy Pain Relief: Randomized Controlled Trial. Surg Laparosc Endosc Percutan Tech. 2017 Aug;27(4):228-232. doi: 10.1097/SLE.0000000000000405. PMID 28472015